CLINICAL TRIAL: NCT01992198
Title: Escalade or Deseacalade Antibiotic Use in Severe Acute Pancreatitis
Brief Title: Multi-center Clinical Study of Early Antibios of Severe Acute Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erzhen Chen (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Sponsor-Investigator, Erzhen Chen, Professer, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAP BUNDLE-ANTIBIOTICS; 12411950500 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2013-10-31; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatitis,Acute Necrotizing
Keywords: antibiothearpy strategy; cefoperazone; metronidazole; meropenem
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing | interventions — Cefoperazone; Metronidazole; chlorhexidine gluconate; Enteral Nutrition; Somatostatin; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cefoperazone + metronidazole (Experimental): cefoperaozone 2g q8h + MDZ 0.5g q8h Oral care Somatostatin 3-6mg per 24h enteral nutrition
  Interventions: Procedure: oral care by chlorhexidine gluconate; Procedure: enteral nutrition; Drug: Somatostatin; Drug: Meropenem
- meropenem (Active Comparator): Meropenem 0.5g q6h or adapted with renal function. Oral care Somatostatin 3-6mg per 24h enteral nutrition
  Interventions: Drug: cefoperazone + metronidazole; Procedure: oral care by chlorhexidine gluconate; Procedure: enteral nutrition; Drug: Somatostatin

INTERVENTIONS:
Drug: cefoperazone + metronidazole — 1.Clinical parameters (2 of 3):
  1)temperature<37.8℃ or 2)HR <100bpm or 3)SpO2 >95% 2.Laboratory parameters (3 of 3):
  1)CRP or 2)PCT reduction 70% compared to zenith for 2 consecutive samples 3)WBC <12×10E9/L for 2 consecutive samples 3.Image parameter (1 of 1): liquid collection developed <30% compared to that of 72h
  Other Names: Cefobid; Metronidazole
  Arms: meropenem
Procedure: oral care by chlorhexidine gluconate — oral care by 0.2% chlorhexidine gluconate twice daily
  Other Names: chlorhexidine gluconate
Procedure: enteral nutrition
  Other Names: Enteral Nutritional Suspension(SP) by NUTRICIA
Drug: Somatostatin
  Other Names: somatostatin by merk
Drug: Meropenem — All patients in cefo-group do not meet 1 of 3 laboratory parameter or image parameter or 2 of 3 clinical parameters.
  1.Clinical parameters (2 of 3):
  1)temperature<37.8℃ or 2)HR <100bpm or 3)SpO2 >95% 2.Laboratory parameters (3 of 3):
  1)CRP or 2)PCT reduction 70% compared to zenith for 2 consecutive samples 3)WBC <12×10E9/L for 2 consecutive samples 3.Image parameter (1 of 1): liquid collection developed <30% compared to that of 72h
  Arms: cefoperazone + metronidazole

SUMMARY:
Strategy of antibiotic therapy in SAP,De-escalate (cefoperazone+metronidazole) or Escalate (meropenem) therapy,which one is better.

DETAILED DESCRIPTION:
SAP is a serious and life-threatening disease and requires intensive and aggressive management of multiple organ failure and severe infectious complications that can develop in these patients. The most common cause of death in patients suffering from severe acute pancreatitis (SAP) is the infection of pancreatic necrosis by enteric bacteria with mortality rates of 30% (range 14- 62%),spurring the discussion of whether or not prophylactic antibiotic administration could be a beneficial approach. Pancreatic infections are more often monomicrobial, especially E. coli in the two first weeks (100% and 62.5%) of onset, with a shift from gram-negative to gram-positive as the pancreatitis progressed.

In order to evaluate the benefit of prophylactic antibiotic application, a number of randomized controlled clinical trials have been published over the past 15 years. Since the results were conflicting and most studies were of low methodological quality and/or statistically underpowered, meta-analyses have been performed to assess this important issue. However, their results ranged from absolutely no effect of antibiotic prophylaxis to positive effects regarding mortality, the incidence of infected pancreatic necrosis and the incidence of extra pancreatic infections.

In order to provide reliable evidence of the effect of antibiotherapy strategy in SAP, we performed a prospective randomized multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* severe Acute Pancreatitis according to Atlanta criteria revisited in 2012

Exclusion Criteria:

* concurrent sepsis or (peri)pancreatic infection caused by a second disease
* patients with chronic organ failure (chronic renal failure needs kidney replacement, chronic heart failure, decompensate hepatic cirrhosis, chronic obstructive pulmonary disease)
* recurrent or endoscopic retrograde cholangiopancreatography (ERCP), or traumatic or operative pancreatitis
* pregnancy, malignancy or immunodeficiency
* a history of allergy to meropenem, cefoperazone and metronidazole
* a history of antibiotic administration within 48 h prior to enrollment
* possible death within 48 h after enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
pancreatic or peripancreatic infection | 28-day

SECONDARY OUTCOMES:
cost of management of SAP | 90-day
Microbiology resistance | 90-day
  sputum, urine and blood culture will be done once or twice per week if needed. bill or other culutre will be done when the patient is undergoing operation.

CONTACTS AND LOCATIONS:
Overall Officials: Er-Zhen Chen, M.D. & Ph.D., Study Chair — Ruijin Hospital; En-Qiang Mao, M.D. & Ph.D., Study Director — Ruijin Hospital; Zhi-Tao Yang, M.D. & Ph.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Depatrment of EICU,Ruijin Hospital, Shanghai, Shanghai Municipality, China